CLINICAL TRIAL: NCT01030471
Title: Supporting Treatment Adherence Needs in Diabetes: The STAND Study
Brief Title: Supporting Treatment Adherence Needs in Diabetes
Acronym: STAND
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: poor accrual
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DK81711; R03DK081711 (NIH)
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2011-06

CONDITIONS: Type 1 Diabetes
Keywords: adolescents; depression; adherence; family functioning; intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: Family-based cognitive-behavioral treatment
- Wait list control group (No Intervention)

INTERVENTIONS:
Behavioral: Family-based cognitive-behavioral treatment — Participants will engage in ten weekly sessions aimed at improving depressive symptoms and medication compliance via reducing family conflict and improving communication among family members.
  Arms: Lifestyle counseling

SUMMARY:
There is an unmet treatment need for depressed adolescents with type 1 diabetes. To address this unmet need, we have designed a new, family-based, cognitive-behavioral intervention to reduce depressive symptoms, improve family functioning, and improve medication compliance. The intervention is delivered in two phases (1 - reduction of depressive symptoms and family conflict, 2 - adherence promotion) as efforts to improve adherence will have a greater likelihood of success if individual and family functioning variables are addressed first. To test the effectiveness of this intervention in reducing depressive symptoms and improving adherence, we will conduct a randomized controlled trial comparing this new intervention to usual care in a sample of fifty-two adolescents with type 1 diabetes and their primary caregivers. Given the absence of this type of intervention and the significance of the problem, this study is timely and important, as it has the potential to positively impact diabetes-specific health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-17
* Diagnosis of type 1 diabetes according to criteria from the ADA for at least 1 year
* Daily insulin dosing of at least 0.5 units per kilogram per day
* Clinical elevation on the CDI (i.e., score at or above 13)
* Assent to participation in study

Exclusion Criteria:

* Other chronic, physical disease or condition except for celiac or thyroid disease
* Diagnosis of major mental disorder (e.g., bipolar disorder, thought disorder, anorexia nervosa)
* Diagnosis of developmental disorder (e.g., mental retardation, autism, Asperger's)
* Current enrollment in psychotherapy specifically targeting depression

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Children's Depression Inventory (CDI)-Measure of adolescent depressive symptoms | Assessed at 0, 1.5, 3, and 6 months after enrollment
Diabetes-Related Family Conflict Scale (DFCS)-Measure of family conflict around diabetes-specific tasks | Assessed at 0, 1.5, 3, and 6 months from enrollment

SECONDARY OUTCOMES:
Hemoglobin A1c value | Obtained at 0, 3, and 6 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Korey K Hood, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States